CLINICAL TRIAL: NCT03136601
Title: Percutaneous Tibial Nerve Stimulation Maintenance: Monthly Therapy or Per Patient Requested Need
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Tajnoos Yazdany, M.D., Physician, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30996-01
Record Dates: First submitted 2017-04-07; First posted 2017-05-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2018-05

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PTNS monthly (Active Comparator): Patients return for PTNS maintenance monthly.
  Interventions: Other: PTNS maintenance
- PTNS as needed (Experimental): Patients return for PTNS as needed (2-12 weeks).
  Interventions: Other: PTNS maintenance

INTERVENTIONS:
Other: PTNS maintenance — The intervention is the timing of PTNS for maintenance (monthly treatment versus as patient needs)

SUMMARY:
The overall objective of this study is to compare the efficacy of the standard monthly maintenance therapy for percutaneous tibial nerve stimulation (PTNS), to sessions as the patient needs (prn) between 2 weeks and 12 weeks, based on overactive bladder symptoms. This is study is to help determine feasibility for conducting a larger trial that is appropriately powered to provide meaningful data.

DETAILED DESCRIPTION:
Patient will be recruited from the Urogynecology clinic on the first floor of the hospital. Patients who have completed 12 weeks of PTNS therapy will be identified by the clinic nurse or nurse practitioner and then a member of the research team will approach the patient regarding involvement in the study. Patients will be asked if they would like to take part in this study and will be given the human bill of rights and well as consent forms in their preferred language (English or Spanish) if they agree to participate. Once they agree to participate, they will be asked to sign the consent forms in a private patient room.

This is a pilot study for feasibility designed as an equivalence and cost analysis study. Patients will be recruited at the 12th session of PTNS (conclusion of treatment and before maintenance therapy starts).

Patients will be from the Urogynecology clinic at Harbor UCLA Medical Center who have OAB and who have been treated with the standard 12 sessions of PTNS. Patients will be randomized to "every month PTNS maintenance" or "as needed PTNS maintenance (Q2-12 weeks)." At enrollment, questions will be read to patients in either Spanish or English based on patient's preferred language and study staff will fill out the surveys for the patient. The patient with the study staff will complete the validated questionnaires, Overactive Bladder Questionnaire (OAB-q), the Benefit, Satisfaction and Willingness to Continue the Treatment questionnaire (BSW) and the Visual analogue scale for satisfaction with treatment. Urinary symptoms will be measured by the validated Overactive Bladder Symptom Scale (OAB-SS) and a modified voiding diary. All patients will have a urine dip completed at this visit to rule out a bladder infection. Finally patients, with the help of study staff, will answer open ended questions. All of these measures will be repeated 3 months after enrollment and one year from enrollment. After the yearlong study, participants can continue treatment which will be decided by the patient and treating clinician. A cost analysis will compare the cost to patients and the cost to the clinic between the monthly PTNS maintenance group and the patient prn maintenance group. All of the above measures will be recorded at enrollment, 3 months from enrollment and 1 year from enrollment. This will be done in person with the help of the study staff at enrollment and either in person, via the phone or in writing at 3 month and 1 year follow up. No payment and no other recruitment methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if they have completed 12 session of PTNS treatment and agree to continue with maintenance therapy.
* Inclusion criteria is Women >=18 years of age, Completed 12 weeks of PTNS and desire to continue,
* Capable of giving informed consent, primary language of English or Spanish,
* Ambulatory and able to use toilet independently without difficulty, Capable and willing to follow all study-related procedures, OAB

Exclusion Criteria:

* Exclusion criteria includes Botox® use in bladder or pelvic floor muscles within past one year,
* Current urinary tract infection, Male, under 18 years old, non-English or Spanish speaking, patients who are unable to consent for themselves, prisoners, pregnant patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Urogynecology clinic setting where only female patients are seen.
Enrollment: 37 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Quality of Life - change | 3 months and 12 months from enrollment
  The primary aim is patient reported quality of life. A validated quality of life questionnaire specific to overactive bladder (OAB) (OAB-q).

SECONDARY OUTCOMES:
Patient Satisfaction- change | 3 months and 12 months from enrollment
  The secondary aim is patient satisfaction which will be measured by the validated questionnaire, Benefit, Satisfaction and Willingness to Continue the Treatment questionnaire (BSW).

OTHER OUTCOMES:
Urinary Symptoms - change | 3 months and 12 months from enrollment
  The tertiary aim is urinary symptoms which will be measured by the validated Overactive Bladder Symptom Scale (OAB-SS).

CONTACTS AND LOCATIONS:
Locations (1):
- Harbor UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No